CLINICAL TRIAL: NCT05967754
Title: Correlation Between Serum Uric Acid and Pulmonary Arterial Hypertension Based on Echo Probability in Patients With Obstructive Sleep Apnea Syndrome
Brief Title: Correlation Between Serum Uric Acid and Pulmonary Hypertension in Obstructive Sleep Apnea Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Rania Ahmad Sweed, clinical professor, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 24/327
Record Dates: First submitted 2023-07-15; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Polysomnography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Obstructive sleep Apnea (Other): Patients with Obstructive sleep Apnea
  Interventions: Diagnostic Test: polysomnography

INTERVENTIONS:
Diagnostic Test: polysomnography — polysomnography and serum uric acid measurement

SUMMARY:
This study aimed to correlate serum uric acid levels and PAH in OSAHS patients.

DETAILED DESCRIPTION:
Obstructive sleep apnea-hypopnea syndrome is the most common form of SRBDs. Recurrent hypoxia, that accompanies OSAHS increases the degradation of ATP, which in turn increase uric acid concentration that can be used as a biomarker of tissue hypoxia in OSAHS. There is still debate about whether OSAHS is an independent contributor to pulmonary arterial hypertension.

AIM OF THE WORK This study aimed to correlate serum uric acid levels and PAH in OSAHS patients. Methods We enrolled 100 patients diagnosed with OSAHS using polysomnography. Patients were divided into three severity groups: mild OSA (5 ≤ AHI < 15), moderate OSA (15 ≤ AHI < 30), and severe (30 ≤ AHI < 60). Serum uric acid was measured the morning after polysomnography. All patients underwent standard echocardiograms, and Pulmonary artery systolic pressure calculation was done.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of OSAHS by overnight polysomnography (AHI ≥ 5/ hr)
* ≥18 years old.

Exclusion Criteria:

* Other sleep disorders as narcolepsy or hypersomnia were excluded as well as Patients with neuropsychiatric disorders.
* Hemodynamically unstable patients
* Patients with other chronic respiratory or cardiac diseases
* Patients with other known causes of pulmonary hypertension
* Patients with any disease or on medication that could alter excretion or urinary metabolism of uric acid such as Excessive uric acid production

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
This study aimed to correlate serum uric acid levels and Pulmonary Arterial Hypertension in Obstructive Sleep Apnea Hypopnea Syndrome patients. | one Year
  This study aimed to correlate serum uric acid levels and Pulmonary Arterial Hypertension in Obstructive Sleep Apnea Hypopnea Syndrome patients.

CONTACTS AND LOCATIONS:
Overall Officials: rania A SEWIED, doctor, Principal Investigator — alex
Locations (1):
- Rania Ahmad Sweed, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No